CLINICAL TRIAL: NCT06192095
Title: Applying Liquid Skin Barrier Film to Prevent Skin Complications Around Indwelling Vascular Catheters in Pediatric Patients: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital Yunlin Branch, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202310113DIND; NTUHYL 113-X015 (Other Grant/Funding Number: National Taiwan University Hospital Yunlin Branch)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Skin Injury; Skin Allergy
Keywords: Indwelling vascular catheters; Liquid skin barrier film; Wound dressing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without skin barrier film (No Intervention): Routine care without skin barrier film around the insertion site of a vascular indwelling catheter
- With skin barrier film (Experimental): Routine care with preventive use of skin barrier film around the insertion site of a vascular indwelling catheter
  Interventions: Device: Skin barrier film

INTERVENTIONS:
Device: Skin barrier film — Preventive use of skin barrier film after insertion of a vascular indwelling catheter before covering with transparent dressing +/- gauze
  Arms: With skin barrier film

SUMMARY:
Long-term indwelling vascular catheters including central venous catheters, peripherally inserted central venous catheters, arterial catheters are often essential for medical care. During the routine care, some patients may experience skin damage around the catheter insertion site due to allergic reactions to the catheter dressing material, physical damage during dressing changes, leading to infection, prolonged hospitalization, and unexpected medical costs. If the condition is mild, it may increase the number of dressing changes. In severe cases, it may require changing to a different dressing method, using medication, or even removing the indwelling catheter. This study investigates the efficacy of liquid skin barrier film in preventing skin damage around long-term indwelling vascular catheters. In this randomized controlled trial, the participants aged 0 to less than 18 years who has long-term indwelling vascular catheters inserted at National Taiwan University Hospital Yunlin Branch will be recruited. At the time of indwelling vascular catheter insertion, the subjects are randomly assigned to the control group or the experimental group. The control group received standard care according to the hospital's guidelines, using a sterile transparent dressing or gauze to cover the catheter insertion site. The experimental group first applied liquid skin barrier film to the skin, then applied a sterile transparent dressing or gauze to cover the catheter insertion site. The patients are followed for two weeks. The primary endpoint is the need for change of dressing, use of medication, or removal of the catheter due to skin damage around the catheter insertion site. The secondary endpoints are skin breakdown, number of dressing changes, and incidence of bloodstream infection. It is expected that the research results may change the standard clinical management of long-term indwelling vascular catheters.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17 years (less than 18 years old)
* Receiving a central venous catheter, peripherally inserted central catheter, or arterial line insertion

Exclusion Criteria:

* The skin around the catheter insertion site is not inact
* Known allergic to liquid skin barrier film

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change of dressing method | 0-14 days
  Change of dressing method due to injury/allergy of skin around the vascular indwelling catheters
Medical treatment for the skin | 0-14 days
  Need of medical treatment (topical, oral, intravenous) due to injury/allergy of skin around the vascular indwelling catheters
Vascular indwelling catheter removal | 0-14 days
  Need of catheter removal due to injury/allergy of skin around

SECONDARY OUTCOMES:
Occurrence of skin injury/allergy | 0-14 days
  Skin injury/allergy of the skin around the vascular indwelling catheter
Pain degree/severity of the skin | 0-14 days
  Pain degree of the skin around the vascular indwelling catheter
Number of dressing changes | 0-14 days
  Total number of dressing changes of the vascular indwelling catheter
Catheter-related bloodstream infection | 0-14 days
  Occurrence of catheter-related bloodstream infection

CONTACTS AND LOCATIONS:
Overall Officials: Hīng-Ka Lîm, MD, PhD, Principal Investigator — National Taiwan University Hospital; Ching-Ching Yang, RN, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: No